CLINICAL TRIAL: NCT06941181
Title: Neurocognitive Predictors of Health Risk Behaviors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Jungmeen Kim-Spoon, Principal Investigator, Virginia Polytechnic Institute and State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Predictors of Risky Behaviors
Record Dates: First submitted 2025-04-14; First posted 2025-04-23 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Substance Use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neurocognition (Other): Neurocognitive tasks
  Interventions: Other: neurocognitive tasks

INTERVENTIONS:
Other: neurocognitive tasks — 1. risk-processing: Participants choose between two choices across 72 trials of a forced choice decision-making neurocognitive task (Holt and Laury, 2002). Each trial included a high and low monetary outcome with an associated probability of occurring. Each choice option is shown as a pie with ten slices represented probabilities, in which each piece corresponded to ten percent.
  2. cognitive control: A multi-source interference task (MSIT; Bush et al., 2003) is used in which participants are presented with three digits and asked to identify the digit different from the others. In the neutral condition, the target's identity is congruent with its relative position. In the interference condition, the target's identity does not match its relative position. There are a total of 96 neutral trials and 96 interference trials.

SUMMARY:
This study proposes to extend the ongoing longitudinal study of health risk behaviors and obtain new data from former adolescents (followed previously from ages 13-22; Times 1-8) now from ages 23 to 28 (Times 9-11). The goal of this study is to examine the contribution of developing neurocognitive markers to substance use in young adulthood by following a well-characterized longitudinal sample.

DETAILED DESCRIPTION:
The main questions it aims to answer is: what are the long-term effects of valuation and control decision-making systems on health risk behaviors? Participants will complete online surveys assessing their substance use behaviors and perform neurocognitive tasks related to risk processing and cognitive control across three time points.

ELIGIBILITY:
Inclusion Criteria:

- Adolescents (now young adults) who participated in the original longitudinal project.

Exclusion Criteria:

* standard contraindications for magnetic resonance imaging at the study onset
* history of seizures/stroke
* a head injury with > 10 min of unconsciousness or neurological sequelae

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2014-01-20 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
substance use behaviors | Approximately every 18 months, 3 times across 5 years
  Frequency (past year and past month use) of cigarette/tobacco, alcohol, cannabis, and other drug use will be asked.

CONTACTS AND LOCATIONS:
Overall Officials: Jungmeen Kim-Spoon, PhD, Principal Investigator — Virginia Polytechnic Institute and State University; Brooks Casas, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (2):
- United States (2):
  - Virginia Tech, Blacksburg, Virginia
  - Fralin Biomedical Research Institute at VTC, Roanoke, Virginia